CLINICAL TRIAL: NCT06164951
Title: A Phase 3, Multicenter, Double-Blind, Randomized, Placebo-Controlled Study to Evaluate the Efficacy and Safety of Infigratinib in Children 3 to <18 Years of Age With Achondroplasia: PROPEL 3
Brief Title: A Study to Evaluate the Efficacy and Safety of Infigratinib in Children and Adolescents With Achondroplasia
Acronym: PROPEL3
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: QED Therapeutics, a BridgeBio company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: QBGJ398-303
Record Dates: First submitted 2023-11-29; First posted 2023-12-11 (Actual); Last update posted 2025-11-12 (Actual); Status verified 2025-11

CONDITIONS: Achondroplasia
Keywords: Skeletal dysplasia; Endochondral ossification; Quality of life in achondroplasia; Fibroblast growth factor receptor 3; FGFR3; Endochondral bone formation; Short-limb disproportionate dwarfism; Dwarfism; Bone disease; Functionality in achondroplasia; Musculoskeletal diseases; Osteochondrodysplasia; Genetic diseases; Long-term treatment; Growth; Annualized height velocity
MeSH Terms: conditions — Achondroplasia; Mucopolysaccharidosis IV; Dwarfism; Bone Diseases; Musculoskeletal Diseases; Osteochondrodysplasias; Genetic Diseases, Inborn | interventions — infigratinib

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Infigratinib 0.25 mg/kg/day (Experimental): Infigratinib at 2, 3.5, 5, 7, 10 mg
  Interventions: Drug: Infigratinib 0.25 mg/kg/day
- Placebo 0.25 mg/kg/day (Placebo Comparator): Placebo Comparator at 2, 3.5, 5, 7, 10 mg
  Interventions: Drug: Placebo Comparator 0.25 mg/kg/day

INTERVENTIONS:
Drug: Infigratinib 0.25 mg/kg/day — Daily doses of oral Infigratinib (sprinkle capsules) at 2, 3.5, 5, 7, 10 mg
  Arms: Infigratinib 0.25 mg/kg/day
Drug: Placebo Comparator 0.25 mg/kg/day — Daily doses of oral Placebo Comparator (sprinkle capsules) at 2, 3.5, 5, 7, 10 mg
  Arms: Placebo 0.25 mg/kg/day

SUMMARY:
This is a Phase 3, multicenter, double-blind, randomized, placebo-controlled study to evaluate the efficacy and safety of infigratinib in children and adolescents with achondroplasia (ACH) who have completed at least 26 weeks of participation in the QED-sponsored study PROPEL (QBGJ398-001).

ELIGIBILITY:
Inclusion Criteria:

1. Subject must be 3 to <18 years of age at screening with growth potential defined as annualized height velocity of >1.5 cm/year over a period of at least 6 months of participation in the PROPEL observational study (QBGJ398-001), pubertal Tanner stage ≤4, and bone age ≤13 years in females and ≤15 years in males.

   Type of Subject and Disease Characteristics
2. Subjects who have a diagnosis of ACH that has been documented clinically and confirmed by genetic testing.
3. Subjects must have completed at least 26 weeks in the PROPEL (QBGJ398-001) study before screening.
4. Subjects are able to swallow oral medication.
5. Subjects and parent(s), legal guardian(s), or caregivers are willing and able to comply with study visits and study procedures.
6. Subjects are ambulatory and able to stand without assistance.

   Sex and Contraceptive/Barrier Requirements
7. Negative pregnancy test in girls ≥10 years of age or girls of any age who have experienced menarche.
8. If sexually active, subjects, whether male or female, must be willing to use a highly effective method of contraception while taking study drug and for 3 months after the last dose of study drug.

   Informed Consent
9. Signed informed consent, which includes compliance with the requirements and restrictions listed in the informed consent form and in this protocol, must be obtained for each subject from their parent(s) or legal guardian and signed informed consent/assent must be obtained from the subject (when applicable)

Exclusion Criteria:

Medical Conditions

1. Subjects who have hypochondroplasia or short stature condition other than ACH.
2. Significant concurrent disease or condition that, in the view of the investigator and/or sponsor, would confound assessment of efficacy or safety of infigratinib.
3. Current evidence of clinically significant corneal or retinal disorder/keratopathy -confirmed by ophthalmic examination.
4. Concurrent circumstance, disease or condition that, in the view of the investigator and/or sponsor, would interfere with study participation or safety evaluations and/or would require treatment with a prohibited medication, and/or would place the subject at high risk for poor treatment compliance or for not completing the study.
5. History and/or current evidence of extensive ectopic tissue calcification.
6. History of malignancy.

   Prior/Concomitant Therapy
7. Having received or planning to receive treatment with any other investigational or approved product for the treatment of ACH or short stature.
8. Regular long-term treatment (≥3 weeks) with supraphysiologic doses of glucocorticoid therapy (ie, >15 mg/m2/day of hydrocortisone or equivalent) or treatment with glucocorticoids at anti-inflammatory doses (ie, 2.5-10 mg/kg/day of hydrocortisone or equivalent) for over 3 weeks within 6 months of the screening visit (low-dose local preparations including inhaled steroid for asthma, intranasal sprays for allergies, and topical steroids are allowed).
9. Previous limb-lengthening surgery at any time or planned/expected to have limb-lengthening surgery or guided growth surgery during the study period. Guided growth surgery with plates removed at least 12 months prior to screening is allowed.
10. Currently receiving treatment with agents that are known strong inducers or inhibitors of CYP3A4 or prolonged treatment (>1 week) with medications that alter the pH of the gastrointestinal tract including antacids, H2 antagonists (eg, ranitidine, famotidine), and proton-pump inhibitors (eg, omeprazole).
11. Current evidence of endocrine alterations of calcium/phosphorus homeostasis.

    Diagnostic assessments
12. Subjects who have significant abnormality in screening laboratory results.

    Other Exclusions
13. Having had a fracture of the long bones (ie, extremities) or spine within 12 months prior to screening.
14. Pregnant or breastfeeding at the screening visit or planning to become pregnant (self or partner) at any time during the study.
15. Allergy or hypersensitivity to any components of the study drug.

Ages: 3 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 110 (Estimated)
Dates: Start 2023-11-10 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-04-30 (Estimated)

PRIMARY OUTCOMES:
Change from baseline (BL) in annualized height velocity (cm/year) | Week 52

SECONDARY OUTCOMES:
Change from BL in height Z-score (in relation to ACH tables) | Week 52
Change from BL in upper to lower body segment ratio | Week 52
Change from BL in height Z-score (in relation to non-ACH tables) | Week 52
Annualized height velocity (cm/year) | Week 52
Absolute and change from baseline in upper arm to forearm length ratio (cm) | Week 52
Absolute and change from baseline in upper leg to lower leg length ratio (cm) | Week 52
Absolute and change from baseline in arm span (cm) to standing height ratio | Week 52
Absolute and change from baseline in head circumference (cm) to standing height ratio | Week 52
Absolute value and change in body mass index | Week 52
Incidence of adverse events | Week 52
Change from BL in annualized height velocity (cm/year) in children 5 years old and older, compared to placebo | Week 52
Change from BL in the Physical Functioning dimension of the Pediatric Quality of Life Generic Core Scale Short Form | Week 52
  Scale scores 0-100. Higher score=better Health-Related Quality of Life
Change in psychomotor function assessed by age-appropriate computerized tests (Detection Test), compared to placebo | Week 52
  Lower score=better performance. Range values=2-6
Change from BL in attention assessed by age-appropriate computerized tests (Identification Test) | Week 52
  Lower score=better performance. Range values=2-6
Change from BL in visual learning assessed by age-appropriate computerized tests (One Card Learning Test) | Week 52
  Higher score=better performance. Range values=0-1.6
Change from BL in working memory assessed by age-appropriate computerized tests (One Back Test) | Week 52
  Lower score=better performance. Range values=2-6
Pharmacokinetic profile of infigratinib by assessment of maximum concentration (Cmax) | Week 52
Pharmacokinetic profile of infigratinib by assessment of time-to-maximum concentration (Tmax) | Week 52
Change from BL in collagen X marker concentration (ug/L) | Week 52
Evaluate the acceptability and palatability of infigratinib using a 5-point hedonic scale | Week 13

CONTACTS AND LOCATIONS:
Overall Officials: QED Therapeutics, Inc. Medical Director, Clinical Development, Study Director — QED Therapeutics
Locations (27):
- United States (7):
  - QED Investigative Site, San Francisco, California
  - QED Investigative Site, Aurora, Colorado
  - QED Investigative Site, Baltimore, Maryland
  - QED Investigative Site, Columbia, Missouri
  - QED Investigative Site, Cincinnati, Ohio
  - QED Investigative Site, Nashville, Tennessee
  - QED Investigative Site, Madison, Wisconsin
- QED Investigative Site, Buenos Aires, Buenos Aires F.D., Argentina
- QED Investigative Site, Parkville, Victoria, Australia
- Canada (4):
  - QED Investigative Site, Edmonton, Alberta
  - QED Investigative Site, London, Ontario
  - QED Investigative Site, Ottawa, Ontario
  - QED Investigative Site, Montreal, Quebec
- France (3):
  - QED Investigative Site, Bron
  - QED Investigative Site, Paris
  - QED Investigative Site, Toulouse
- QED Investigative Site, Rome, Italy
- Norway (2):
  - QED Investigative Site, Bergen
  - QED Investigative Site, Oslo
- QED Investigative Site, Singapore, Singapore
- Spain (2):
  - QED Investigative Site, Málaga
  - QED Investigative Site, Vitoria-Gasteiz
- United Kingdom (5):
  - QED Investigative Site, Bristol
  - QED Investigative Site, Glasgow
  - QED Investigative Site, London
  - QED Investigative Site, Manchester
  - QED Investigative Site, Sheffield

IPD SHARING:
Plan to Share IPD: No